CLINICAL TRIAL: NCT03750773
Title: GRIPP: Gabapentin for Relief of Immediate Postoperative Pain
Brief Title: Gabapentin for Relief of Immediate Postoperative Pain
Acronym: GRIPP
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, David Haas, Robert A. Munsick Professor of Obstetrics and Gynecology with Tenure, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1809661339
Record Dates: First submitted 2018-11-16; First posted 2018-11-23 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Randomized 1:1 drug:placebo in blocks of 6 stratified by the hospital, double blind study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Subjects receiving gabapentin drug (Active Comparator): Administration of Gabapentin 600mg orally every 8 hours. Women will receive gabapentin for a total of 48 hours after cesarean
  Interventions: Drug: Gabapentin 600mg
- Subjects receiving placebo oral capsule (Placebo Comparator): Administration of identical placebo capsule orally every 8 hours. Women will receive placebo for 48 hours after cesarean
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Gabapentin 600mg — Subject is given Gabapentin 600mg every 8 hours x 48 hours postoperatively for pain control.
  Arms: Subjects receiving gabapentin drug
Drug: Placebo oral capsule — Subject is given a Placebo capsule every 8 hours x 48 hours postoperatively for pain control.
  Arms: Subjects receiving placebo oral capsule

SUMMARY:
The purpose of this study is to use gabapentin as an additional or alternative treatment for short term pain control following cesarean delivery in order to reduce the use of opioid pain medication and improve overall pain control following surgery.

DETAILED DESCRIPTION:
This is a randomized, placebo controlled, double blind study. After consent, the subject will complete a Depression Screening to establish a baseline score. Within 2 hours following completion of a cesarean section, the subject will be given the study drug (600mg Gabapentin) or placebo. She will be given this every 8 hours for 48 hours scheduled. She will also have the option to take routine opioid pain medication if her pain is uncontrolled. She will be asked to rate her postoperative pain on a Visual Analog Scale prior to receiving the study drug, 2-4 hours after each dose, and at 24, 36, and 48 hours postoperatively. For breastfeeding infants, data will be collected regarding overall feeding quality, somnolence levels, gestational age at birth, infant weight at birth and discharge, the highest bilirubin level while inpatient and any treatment for this as applicable. The subject will complete the Depression Scale again at 48 hours following delivery. At one week postpartum, they will receive a phone call and the following will be addressed: a final pain survey, a Depression survey, nausea level, number of pain pills left in their prescription, adverse events, whether or not they would take the study drug again if they should happen to have another cesarean section, and infant well-being if breastfeeding.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women at least 18 years of age
2. Gestational age > or = to 30 weeks
3. Singleton gestation
4. Women undergoing a non-emergent cesarean delivery
5. Spinal anesthesia or combined spinal-epidural anesthesia utilized during cesarean
6. Ability to undergo the informed consent process in English

Exclusion Criteria:

1. Vertical skin incision
2. General anesthesia for cesarean
3. History of major depression or postpartum depression requiring medication
4. Chronic opiate use during pregnancy, defined as anyone who has taken an opioid or opioid replacement therapy in the 3 days prior to admission for delivery. This does not include opioids given for labor anesthesia.
5. Magnesium sulfate treatment postpartum
6. Preexisting fibromyalgia, chronic pain syndrome, or rheumatologic disorder

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07-02 (Estimated); Primary Completion 2020-03 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Total morphine milligram equivalents consumed in the first 48 hours postoperatively | 48 hours
  The total morphine milligram equivalents consumed by the subjects within the first 48 hours postoperatively will be recorded and compared between the two arms.

SECONDARY OUTCOMES:
Total morphine milligram equivalents from hospital discharge to one week postoperatively | one week
  The total number of pills of postoperative opioid pain medication consumed will be recorded, converted into morphine milligram equivalents, and compared between the two arms.
Subject reported pain rating on a Visual Analog Scale within the first 48 hours postoperatively | 48 hours
  Each subject will report a measure of pain on a Visual Analog Scale before and 2-4 hours after each dose of study drug or placebo, and at 24, 36, and 48 hours postoperatively.
Number and type of adverse events potentially associated with study drug (Safety and Tolerability) | one week
  Adverse events of maternal dizziness, nausea, notable peripheral edema, suicidal behavior or ideation, infant somnolence, and drug reactions will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: David M Haas, MD, MS, Principal Investigator — IUSM, Dept OBGYN

IPD SHARING:
Plan to Share IPD: No